CLINICAL TRIAL: NCT05890976
Title: Efficacy and Safety of Oral Semaglutide 50 mg Once Daily in Chinese Adults With Overweight or Obesity (OASIS 3)
Brief Title: Research Study Looking at How Well Semaglutide Tablets Taken Once Daily Work in Chinese Adults Who Are Above a Healthy Weight Range (OASIS 3)
Acronym: OASIS 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9932-4861; U1111-1266-2400 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide 50 mg (Experimental): Participants will receive semaglutide tablets orally once daily. Participants will receive semaglutide in a dose escalation manner for 44 weeks: 3 mg (weeks 0 to 4), 7 mg (weeks 5 to 8), 14 mg (weeks 9 to 12), 25 mg (weeks 13 to 16) and 50 mg (weeks 17 to 44).
  Interventions: Drug: Semaglutide
- Semaglutide Placebo (Placebo Comparator): Participants will receive placebo tablets matched to semaglutide orally once daily for 44 weeks.
  Interventions: Drug: Semaglutide Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide tablets orally once daily for 44 weeks.
  Arms: Semaglutide 50 mg
Drug: Semaglutide Placebo — Participants will receive placebo matched to semaglutide.
  Arms: Semaglutide Placebo

SUMMARY:
This study is being conducted to see if semaglutide tablets can be used as a treatment to help people who are above a healthy weight range to lose weight. Semaglutide tablets are a new medicine being tested to treat people living with excess body weight. Participants will either get semaglutide or placebo once daily morning for 44 weeks.

In addition to taking the medicine, participants will have talks with study staff about:

* Healthy food choices
* How to be more physically active
* What participants can do to lose weight This study will last for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age greater than or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) of

  1. greater than or equal to 28.0 kilogram per meter square (kg/m^2) or
  2. greater than or equal to 24.0 kg/m^2 with greater than or equal to 1 weight-related comorbidity (treated or untreated). Weight-related comorbidities should be hypertension, T2D, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

For participants with T2D at screening the following inclusion criteria apply in addition to criteria 1- 4:

* Diagnosed with T2D greater than or equal to 180 days prior to screening.
* Treated with either diet and exercise alone or stable treatment (same drug(s) or active ingredient, dose and dosing frequency) for at least 60 days prior to the day of screening with up to 3 oral antidiabetic drugs (OAD)s alone or in any combination (metformin, α-glucosidase (AGI), sulphonylureas (SU), glinides, SGLT2i (sodium-glucose co-transporter 2 inhibitor) or glitazone).
* HbA1c 7.0 - 10.0 percent (53 - 86 millimoles per mole [mmol/mol]) (both inclusive) as measured by central laboratory at screening.

Exclusion Criteria:

Participants without T2D at screening:

* HbA1c greater than or equal to 6.5 percent (48 mmol/mol) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes.
* Treatment with glucose-lowering agent(s) within 90 days prior to screening.

Participants with T2D at screening:

* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of lesser than 30 milli litre per min/1.73 square metre (mL/min/1.73 m^2) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation as defined by Kidney Disease Improving Global Outcomes (KDIGO) 2012 classification by the central laboratory at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Relative Change in Body Weight | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 5 Percent | At end of treatment (week 44)
  Measured as count of participants

SECONDARY OUTCOMES:
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 10 Percent | At end of treatment (week 44)
  Measured as count of participants
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 15 Percent | At end of treatment (week 44)
  Measured as count of participants
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 20 Percent | At end of treatment (week 44)
  Measured as count of participants
Change in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite- CT) - Physical Function Domain | From baseline (week 0) to end of treatment (week 44)
  IWQOL-Lite-CT is a 20-item obesity-specific PRO measure used to assess the impact of body weight changes on patient's physical and psychosocial functioning in three composite scores (Physical Function, Physical and Psychosocial) and a Total score.
Change in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite- CT) - Total score | From baseline (week 0) to end of treatment (week 44)
  IWQOL-Lite-CT is a 20-item obesity-specific PRO measure used to assess the impact of body weight changes on patient's physical and psychosocial functioning in three composite scores (Physical Function, Physical and Psychosocial) and a Total score.
Change in Impact of Weight on Daily Activities Quesionnaire (IWDAQ) - Total Score | From randomisation (week 0) to end-of-treatment (week 44)
  IWDAQ is a 18-item obesity-specific PRO measure developed to evaluate daily activity limitations associated with excess weight. It uses an adaptive questionnaire design where the participant chooses the three IWDAQ activities they would most like to improve with weight loss and rate the degree of limitations in each of the three activities at baseline. The same three activities are assessed for degree of limitations at follow-up to allow for tracking of activities relevant to each individual.
Change in Body Mass Index (BMI) | From baseline (week 0) to end of treatment (week 44)
  Measured in kilogram per square meter (kg/m^2)
Change in Waist Circumference | From baseline (week 0) to end of treatment (week 44)
  Measured in centimeter (cm)
Change in Systolic Blood Pressure | From baseline (week 0) to end of treatment (week 44)
  Measured in millimeter of mercury (mmHg)
Change in Diastolic Blood Pressure | From randomisation (week 0) to end of treatment (week 44)
  Measured in mmHg
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage point (%-point)
Change in Fasting Plasma Glucose | From baseline (week 0) to end of treatment (week 44)
  Measured as milligrams per decilitre (mg/dL)
Change in Fasting Serum Insulin | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in Total Cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in High-density Lipoprotein (HDL) Cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in Low-density Lipoproteins (LDL) Cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in Very Low-density Lipoproteins (VLDL) Cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in Triglycerides | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in Free Fatty Acids | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in High Sensitivity C-reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 44)
  Measured as ratio to baseline
Change in waist-height ratio (WtHR) | From baseline (week 0) to end of treatment (week 44)
Number of Treatment Emergent Adverse Events(TEAE's) | From baseline (week 0) to end of treatment (week 44)
  Measured as count of events
Number of Treatment Emergent Serious Adverse Events(TESAE's) | From baseline (week 0) to end of study (week 51)
  Measured as count of events
AUC 0-24h,sema,50mg,ss: Area Under The Semaglutide-Time Curve (0-24h) During a Dosing Interval at Steady State | Week 20
  Measured as hours*nanomoles per litre (h*nmol/L)
Cmax,sema,50mg,ss: Maximum Concentration at Steady State of Semaglutide 50 mg | Week 20
  Measured as nanomoles per litre (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (16):
- China (16):
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - Huaihe Hospital of Henan University-Endocrinology, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Taihe Hospital-Endocrinology, Shiyan, Hubei
  - The First People's Hospital of Changde City-Endocrinology, Changde, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'nan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Huashan Hospital Fudan University-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com